CLINICAL TRIAL: NCT01227044
Title: Reducing Heavy Drinking to Optimize HIV/AIDS Treatment and Prevention
Acronym: DAWN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0909005730; 1R01AA018923 (NIH)
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Reduction in Heavy Drinking in Patients With HIV
Keywords: Substance Abuse Counseling; Adherence (medication); Alcohol Abuse; Highly Active Antiretroviral Therapy (HAART); Naltrexone; Vivitrol; HIV
MeSH Terms: conditions — Medication Adherence; Alcoholism | interventions — Naltrexone; vivitrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NTX + MM/MC (Active Comparator): Naltrexone + Medical Management/Medication Coaching
  Interventions: Drug: Naltrexone
- Placebo + MM/MC (Placebo Comparator): Placebo plus Medical Management/Medication Coaching
  Interventions: Other: Placebo + Medication Management/Medication Coaching

INTERVENTIONS:
Drug: Naltrexone — NTX arm will receive monthly extended release NTX doses at 380mg (4 mL), administered as an intramuscular gluteal injection at 4-week intervals.
  Other Names: Vivitrol
  Arms: NTX + MM/MC
Other: Placebo + Medication Management/Medication Coaching — Placebo + Medication Management/Medication Coaching
  Arms: Placebo + MM/MC

SUMMARY:
This is a double-blind placebo-controlled study to evaluate the effect of Naltrexone (NTX) and counseling on highly active antiretroviral treatment (HAART) medication adherence in a cohort of HIV-infected patients who report heavy drinking, or meet criteria for alcohol abuse and/or dependence, and inadequate (< 95%) HAART adherence. All patients will receive a behavioral intervention, termed Medical Management/Medication Coaching or MM/MC. MM/MC incorporates the behavioral platform Medical Management (MM) from the National Institute on Alcohol Abuse and Alcoholism (NIAAA)-funded COMBINE Study to reduce heavy alcohol use with Medication Coaching (MC), a manualized treatment designed to improve HAART medication adherence in HIV-infected patients with substance use disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Be HIV-infected.
2. Currently be prescribed HAART medication or be eligible to receive HAART medication.
3. Report less than 95% adherence to their HAART medication.
4. Report heavy drinking 4 or more times in the past 4 weeks, or meet current criteria for alcohol abuse or dependence. Heavy drinking is defined as 4 or more drinks for women and 5 or more drinks for men on one occasion.
5. Be at least 18 years old.
6. Be able to understand English and provide informed consent.

Exclusion Criteria:

1. Be psychotic or severely psychiatrically disabled.
2. Be currently enrolled in formal treatment for alcohol (excluding self-help, e.g. Alcoholics Anonymous)
3. Have medical conditions that would preclude completing or be of harm during the course of the study.
4. Have laboratory or clinical evidence of significant liver dysfunction (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 5 times the upper limit of the normal range) or cirrhosis with a Child-Pugh classification greater than A or B.
5. Have a known contraindication to NTX therapy (e.g. requiring opioid medication for pain).
6. Be pregnant, nursing or unable to use an effective method of birth control (women).

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-04; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E Sullivan (Fiellin), MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University School of Medicine, New Haven, Connecticut
  - VACT Healthcare System, New Haven, Connecticut

REFERENCES:
- [Background] Edelman EJ, Moore BA, Holt SR, Hansen N, Kyriakides TC, Virata M, Brown ST, Justice AC, Bryant KJ, Fiellin DA, Fiellin LE. Efficacy of Extended-Release Naltrexone on HIV-Related and Drinking Outcomes Among HIV-Positive Patients: A Randomized-Controlled Trial. AIDS Behav. 2019 Jan;23(1):211-221. doi: 10.1007/s10461-018-2241-z. PMID 30073637

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NTX + MM/MC | Placebo + MM/MC
Started | 25 | 26
Completed | 19 | 17
Not Completed | 6 | 9
Not completed — Lost to Follow-up | 5 | 7
Not completed — Discontinued Intervention | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + MM/MC | NTX + MM/MC | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (9.2) | 51.2 (7.6) | 51.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 19 | 17 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-non-Hispanic | 2 | 6 | 8
  Black-non-Hispanic | 19 | 17 | 36
  Hispanic | 3 | 1 | 4
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51
ART Adherence [Mean (Standard Deviation); unit: proportion of days adherent] — Presented are the average proportion of days (out of 30) that each participant was ART adherent.
  proportion of days adherent | .59 (.31) | .51 (.33) | .55 (.32)
Undetectable HIV Viral Load [Count of Participants; unit: Participants] | 16 | 10 | 26
CD4 count [Mean (Standard Deviation); unit: cells/mm3] | 513 (423) | 457 (313) | 487 (374)
VACS Score [Mean (Standard Deviation); unit: units on a scale] — The Veterans Aging Cohort Study Index (VACS Index) creates a score by summing pre-assigned points for age, routinely monitored indicators of HIV disease (CD4 count and HIV-1 RNA), and general indicators of organ system injury including hemoglobin, platelets, aspartate and alanine transaminase (AST and ALT), creatinine, and viral hepatitis C infection (HCV) . The potential range is 0-164. A 5 point increase is associated with 20% increased risk of death.
  units on a scale | 44 (26) | 42 (26) | 43 (26)
Heavy Drinking Days in past 30 Days [Mean (Standard Deviation); unit: days] | 16.4 (8.4) | 11.3 (8.4) | 14.7 (9.8)
ANY Drinking Days in past 30 Days [Mean (Standard Deviation); unit: days] | 19.2 (7.5) | 14.8 (8.7) | 17.9 (8.8)
Alcohol Abuse/Dependence [Count of Participants; unit: Participants] | 17 | 18 | 35
Drug Abuse/Dependence [Count of Participants; unit: Participants] | 19 | 20 | 39
Prior Alcohol or Drug Treatment [Count of Participants; unit: Participants] | 15 | 17 | 32
Prior Receipt for Medications to Help with Drinking [Count of Participants; unit: Participants]
  Overall | 3 | 3 | 6
  Naltrexone | 2 | 0 | 2
  Acamprosate | 0 | 1 | 1
  Disulfiram | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: HAART Adherence
Description: The intent of this outcome is to compare the efficacy of NTX +MM/MC versus placebo +MM/MC on adherence to HAART. It is hypothesized that NTX +MM/MC will lead to improved adherence to HAART when compared to placebo + MM/MC.
Time Frame: One year
Population: data were analyzed intention to treat where all observations were included in the analyses, including those only measured at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + MM/MC | NTX + MM/MC
Number analyzed (Participants) | 26 | 25
Participants
  12 Weeks: number analyzed (Participants) | 19 | 16
  12 Weeks | 7 | 4
  24 Weeks: number analyzed (Participants) | 19 | 17
  24 Weeks | 6 | 4
  36 Weeks: number analyzed (Participants) | 19 | 17
  36 Weeks | 8 | 4
  52 Weeks: number analyzed (Participants) | 16 | 13
  52 Weeks | 6 | 3

2. Secondary Outcome: Heavy Drinking Days
Description: This outcome is intended to compare the efficacy of NTX +MM/MC versus placebo +MM/MC in reducing days of heavy drinking. It is hypothesized that NTX +MM/MC will lead to greater reductions in the number of days of heavy drinking when compared to placebo + MM/MC.
Time Frame: One year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo + MM/MC | NTX + MM/MC
Number analyzed (Participants) | 26 | 25
days
  12 Weeks: number analyzed (Participants) | 21 | 19
  12 Weeks | 8.4 (6.8) | 1.7 (4.7)
  24 Weeks: number analyzed (Participants) | 15 | 14
  24 Weeks | 5.4 (8.4) | 0.1 (5.3)
  36 Weeks: number analyzed (Participants) | 16 | 11
  36 Weeks | 4.2 (5.0) | 0.5 (2.0)
  52 Weeks: number analyzed (Participants) | 13 | 9
  52 Weeks | 5.8 (8.3) | 0.3 (4.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected up through the 1 year follow up period.
Arm/Group | Placebo + MM/MC | NTX + MM/MC
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 3/26 | 6/25
Other Adverse Events (participants affected / at risk) | 4/26 | 3/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + MM/MC (N=26) | NTX + MM/MC (N=25)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Intoxication (General disorders) | 3 (6) | 0 (0) — Hospitalization as a result of relapse or intoxication
Suicidal Thoughts (Psychiatric disorders) | 1 (1) | 0 (0)
Testicular Inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 2 (2)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 1 (2)
Hand Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Foot Infection (Infections and infestations) | 0 (0) | 1 (1)
Spinal Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood Clot (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + MM/MC (N=26) | NTX + MM/MC (N=25)
Fall Related Injury (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT01227044/Prot_SAP_000.pdf